CLINICAL TRIAL: NCT06601816
Title: Comparison of Sinus Lifting Techniques Performed with Piezosurgery and a Surgical Guide, a Specially Designed Drill, and Conventional Drills in Terms Complications and Quality of Life
Brief Title: Maxillary Sinus Elevation and Perioperative Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Mehmet Melih Omezli, Professor, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-2323; 23-AKD-48 (Other: Turkish Medicines and Medical Devices Agency)
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Maxillary Sinus Augmentation
Keywords: Sinus floor augmentation; computer-aided design; piezosurgery

STUDY DESIGN:
Intervention Model Description: The three methods used to lift the sinuses were randomized: piezosurgery using a surgical guide, a drill specifically made for lateral sinus lift, and traditional drills.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Reamer Group (Active Comparator): The group in which the lateral window was created with conventional rotary instrument burs
  Interventions: Procedure: maxillary sinus lift with reamer
- Piezo surgery with Surgical Guide Group (Active Comparator): The group in which the lateral window was created using piezo surgery and surgical guide
  Interventions: Procedure: maxillary sinus lift with piezzo
- Conventional Group (Active Comparator): The group in which the lateral window was created with conventional rotary instrument burs
  Interventions: Procedure: maxillary sinus lift with conventional burr

INTERVENTIONS:
Procedure: maxillary sinus lift with reamer — Lateral window created with specially designed burs for lateral sinus lift
  Arms: Reamer Group
Procedure: maxillary sinus lift with piezzo — lateral window was created using piezo surgery and surgical guide
  Arms: Piezo surgery with Surgical Guide Group
Procedure: maxillary sinus lift with conventional burr — the lateral window was created with conventional rotary instrument burs
  Arms: Conventional Group

SUMMARY:
This study aims to investigate the effects of various external sinus lifting techniques on patient comfort and perioperative complications.

DETAILED DESCRIPTION:
Patients who met the inclusion criteria and were admitted for posterior maxilla rehabilitation participated in this prospective, randomized, controlled clinical trial. The three methods used to lift the sinuses were randomized: piezosurgery using a surgical guide, a drill specifically made for lateral sinus lift, and traditional drills. Recorded were the duration of the procedure, accessibility, and intraoperative complications. During the first week following surgery, analgesic intake and pain using a visual analog scale (VAS) were assessed assessed. Preoperatively and on the second and seventh postoperative days, edema was assessed. Preoperatively and on the seventh postoperative day, the patient's quality of life using the OHIP-14 questionnaire, experiences, and expectations were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Severe resorption or sinus pneumatization in the posterior maxilla that prevents standard implant treatment; class V or VI according to Cawood and Howell classification, patients with residual bone height less than 6 mm
2. Patients over 18 years of age
3. Patients without a history of reconstructive pre-prosthetic surgery or previous implant surgery
4. Patients with partial edentulism who have applied to our center for implant treatment and need sinus lifting
5. Patients with cone beam computed tomography (CBCT) taken within the last 1 month

Exclusion Criteria:

1. Patients with a history of systemic diseases (hematologic, neurologic, etc.) that may be contraindicated surgery
2. Patients who are pregnant or in lactation period
3. Patients with a history of immune system disorders and substance abuse
4. Patients with a history of radiotherapy in the head and neck region
5. Patients with existing maxillary sinus pathology or who have undergone surgery
6. Patients who smoke >10 cigarettes per day
7. Patients using antibiotics or steroids in the 30 days before surgery
8. Uncooperative patients who do not comply with the study protocol or follow-up regimen
9. Patients with perforation of the Schneiderian membrane

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Operation Time | from the osteotomy of the sinus window to completation of membrane elevation
  The time from the osteotomy of the sinus window to completation of membrane elevation

SECONDARY OUTCOMES:
Patient Experience | 7th postoperative day
  Patients asked to rate their postoperative experience with a 3-point scale (0, my expectation and experience were the same/similar; 1, my experience was better than my expectation; 2, my experience was worse than my expectation)
Pain | from 6 hours to postoperative 7 days
  intensity of pain experienced by patients assessed using a 10-cm Visual Analogue Scale (VAS)
Analgesic Consumption | from 6 hours to 7 days postoperatively
  need for analgesics
Edema | on the 2nd and 7th days
  Swelling after surgery measurements collected of a anatomical locations on the face that served as reference points. Reference points included the tragus, alare, lateral corner of the eye, gonion, soft tissue pogonion, and external corner of the mouth. The average of each measurement was used to calculate the edema level.
Quality of Life | preoperatively and on postoperative day 7
  The OHIP-14 used to measure quality of life. Scores ranged from 0 (no impact) to 56 (all oral health concerns encountered extremely frequently). It was scored as follows: Never (0 points); Seldom (1 point); Sometimes (2 points); Frequently (3 points); and Very frequently (4 points).
Surgeon;s Comfort | Immediately after surgery
  The comfort of the access to the operation site evaluated by the surgeon on a 4-point scale (0, very poor visibility; 1, fair visibility; 2, good visibility; 3, excellent visibility)

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Ordu, Altınordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozyalcin MS, Omezli MM, Torul D. Effects of Different External Sinus Lifting Techniques on Perioperative Complications and Patient Comfort. Clin Implant Dent Relat Res. 2025 Jun;27(3):e70044. doi: 10.1111/cid.70044. PMID 40320286